CLINICAL TRIAL: NCT03898323
Title: Alcohol Approach Bias Modification Effects on Alcohol Consumption: A Pilot Human Laboratory Study
Brief Title: Pilot Human Laboratory Study of Alcohol Approach Bias Modification (AABM) for Alcohol Use Disorder (AUD)
Acronym: ADP + AABM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: San Francisco VA Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCSF REAC RAP
Record Dates: First submitted 2019-01-02; First posted 2019-04-01 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-05

CONDITIONS: Alcohol Use Disorder
Keywords: human laboratory; alcohol approach bias modification; alcohol use disorder; non-treatment seeking
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- AABM Training (Experimental): Alcohol Approach Bias Modification (AABM) training is a computer training program that participants interact with by pushing and pulling a joystick. Participants are asked to respond to the format of a presented picture, irrespective of the pictures' content. Training effect is achieved by presenting alcohol pictures in push format only and non-alcoholic drinks in pull format only. AABM training consists of 3 sessions per week over 2 weeks, for a total of 6 sessions.
  Interventions: Device: Alcohol Approach Bias Modification

INTERVENTIONS:
Device: Alcohol Approach Bias Modification — Computerized training

SUMMARY:
The overall goal of the proposed project is to improve the treatment of individuals with Alcohol Use Disorder (AUD). We will conduct a pilot feasibility trial of Approach Bias Modification (AABM) training of heavy-drinking non-treatment seeking individuals with AUD. We will measure feasibility with respect to recruitment, retention and tolerability of AABM training and the Alcohol Drinking Paradigm (ADP). We will also assess changes in alcohol craving and alcohol consumption during ADP sessions conducted before and after 2 weeks of AABM training.

DETAILED DESCRIPTION:
Heavy-drinking non-treatment seeking male community volunteers with a diagnosis of AUD will receive 2 weeks of AABM training preceded and followed by a 1-day ADP session.

AABM training is a computer training program that participants interact with by pushing and pulling a joystick. Participants are asked to respond to the format of a presented picture, irrespective of the pictures' content. Training effect is achieved by presenting alcohol pictures in push format only and non-alcoholic drinks in pull format only. Training is conducted in 3 sessions per week for 2 weeks, for a total of 6 sessions.

The ADP session is a one day human laboratory session taking place at the SFVA Medical Center. This human laboratory session involves the self-administration of alcoholic beverages by research participants under highly structured, observed conditions in order to evaluate the effects of the study intervention (AABM training) on alcohol craving and alcohol consumption.

The investigators hoped to recruit 12 participants to enroll and start the clinical trial over the course of 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Men, ages 21-50;
2. Able to read English and to complete study evaluations;
3. Risky (also known as high-risk, or hazardous, or heavy) alcohol use, defined as 25-70 standard drinks per week on average over the past 30 days; Heavy (also known as risky, high-risk, or hazardous) alcohol use, defined as 15-70 standard drinks per week on average over the past 30 days.
4. No more than 3 days/week of alcohol abstinence in the past 30 days, to maximize likelihood that participants will choose to drink during the laboratory sessions.
5. At least 1 heavy drinking day (> 5 drinks/day) per week on average during the 30 days prior to screening.

Exclusion Criteria:

1. Individuals who are seeking AUD treatment or have been in treatment within the past 6 months;
2. Current DSM-V non-alcohol use disorder other than tobacco and marijuana;
3. Positive urine drug test results at more than one baseline appointment for opioids, cocaine, benzodiazepines, or barbiturates;
4. Regular use of psychoactive drugs including antipsychotics, anxiolytics and antidepressants during the 30 days prior to entry, as well as anticonvulsants, beta blockers, central nervous system stimulants or depressants, or other drugs that cause excessive sedation;
5. Psychosis or any other serious mental illness as judged by SCID and study physician assessment;
6. Medical conditions that in the judgment of the study physician contraindicate the consumption of alcohol or would make study participation hazardous;
7. History of serious alcohol withdrawal (e.g. seizures, DTs, hospitalization) or a Clinical Institute Withdrawal Assessment Scale (CIWA-AD) score > 8;
8. Participants who report disliking beer will be excluded because beer will be provided during the alcohol self-administration periods;
9. Participants who have taken any investigational drug within 4 weeks preceding study entry.

Ages: 21 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 3 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven L. Batki, MD, Principal Investigator — University of California, San Francisco/San Francisco VA Health Care System
Locations (1):
- San Francisco VA Health Care System, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AABM Training
Started | 3
Completed | 2
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | AABM Training
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Feasibility
Description: The number of participants who enrolled and actually started study treatment over the 12-month recruitment period.
Time Frame: 12 months
Population: The analysis population consists of the target number (12) of participants that the investigators hoped to recruit and start on study treatment over a 12-month period. There appears to be an inconsistency only because the actual number of participants recruited and started on study treatment over the 12-month period was only 3.
Measure: Count of Participants; unit: Participants
Arm/Group | AABM Training
Number analyzed (Participants) | 12
Participants | 3

2. Primary Outcome: Retention Feasibility
Description: Retention feasibility as measured by the percentage of participants completing Alcohol Drinking Paradigm (ADP) sessions 1 and 2 and completing the 2-week course of 6 AABM training sessions.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AABM Training
Number analyzed (Participants) | 3
Participants | 2

3. Primary Outcome: Tolerability Feasibility
Description: Tolerability feasibility is measured by the number and percent of participants experiencing each adverse event.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | AABM Training
Number analyzed (Participants) | 3
Participants
  Head tingling | 1
  Physically slow | 1
  Sleepiness | 2
  Dizziness | 1
  Itchy/red eyes | 1

4. Secondary Outcome: Alcohol Craving
Description: Alcohol craving will be measured during ADP sessions 1 and 2 using the Alcohol Urge Questionnaire (AUQ).
  Alcohol craving will be measured during Alcohol Drinking Paradigm (ADP) sessions 1 and 2, using the total score of the Alcohol Urge Questionnaire (AUQ). The AUQ has 8 items. Each item is scored on a 1 to 7 scale (Strongly Disagree = 1 and Strongly Agree = 7; items 2 and 7 are reverse scored). Higher scores reflect greater craving. Total score range is from a minimum of 8 to a maximum of 56. The AUQ is administered before alcohol administration and at various times after alcohol administration. The AUQ score reported here is the highest AUQ score obtained for that ADP session.
Time Frame: 6 weeks
Population: One participant did not complete the either ADP session.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | AABM Training
Number analyzed (Participants) | 2
score on a scale
  ADP 1 | 27.3 (6.3)
  ADP 2 | 23.3 (2.6)

5. Secondary Outcome: Alcohol Consumption (Number of Standard Drinks Consumed)
Description: Alcohol consumption will be measured during ADP sessions 1 and 2 using the number of alcoholic standard drinks consumed during ADP session 1 (before 2 weeks of AABM training) and ADP session 2 (after the 2 weeks of AABM training). Consumption was measured using the number of alcoholic standard drinks consumed during the ADP sessions. A standard drink per NIAAA definition is 14 grams of pure alcohol.
Time Frame: 2 days (1 day each for ADP session 1 and 2)
Population: One participant did not complete the either ADP session.
Measure: Mean (Standard Deviation); unit: standard drinks
Arm/Group | AABM Training
Number analyzed (Participants) | 2
standard drinks
  ADP 1 | 1.5 (2.12)
  ADP 2 | 0.5 (0.71)

ADVERSE EVENTS:
Time Frame: Beginning at baseline through the follow-up visit, for a total of 6 weeks.
Groups:
- AABM Training With ADP Sessions Before and After Training: Alcohol Approach Bias Modification (AABM) training is a computer training program that participants interact with by pushing and pulling a joystick. Participants are asked to respond to the format of a presented picture, irrespective of the pictures' content. Training effect is achieved by presenting alcohol pictures in push format only and non-alcoholic drinks in pull format only. AABM training consists of 3 sessions per week over 2 weeks, for a total of 6 sessions.
  Alcohol Approach Bias Modification: Computerized training
Arm/Group | AABM Training With ADP Sessions Before and After Training
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 2/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AABM Training With ADP Sessions Before and After Training (N=3)
Head tingling (Nervous system disorders) | 1 (1)
Physically slow (General disorders) | 1 (1)
Sleepiness/tiredness (General disorders) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1)
Itchy/red eyes (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Of the 3 participants who were assigned to study treatment and who actually started study treatment, 1 participant was withdrawn from the study after ADP session 1. The reason for the study withdrawal was because of study physician decision, based on laboratory test evidence of substance use, making the participant ineligible for study continuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT03898323/Prot_SAP_ICF_001.pdf